CLINICAL TRIAL: NCT00926107
Title: Study of the mTOR Inhibitor Temsirolimus(CCI-779) in Patients With CA125 Only Relapse of Ovarian Cancer. A Phase II Study by the Hellenic Cooperative Oncology Group.
Brief Title: Study of the mTOR Inhibitor Temsirolimus (CCI-779) to Treat Ovarian Cancer With CA125 Only Relapse
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study ended prematurely due to the low accrual rate (24% of the expected accrual rate) in the first two years of patients enrolment
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 4/09; 2008-007925-38 (EudraCT Number)
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus 25mg weekly until clinical progression

SUMMARY:
The primary objective of this study is to determine the efficacy of Temsirolimus in patients with ovarian cancer with CA125 only relapse after first-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof of epithelial ovarian,fallopian or peritoneal carcinoma of the following histological types:serous, endometrioid, mucinous, clear cell, low differentiation.
2. Age 18 years or older
3. Patients should have received first-line platinum based chemotherapy
4. Documented CA125 progression according to GCIC criteria.
5. No evidence of measurable or evaluable disease.
6. Provision of written informed consent
7. ECOG PS 0-2
8. Life expectancy of greater than 12 weeks
9. WBC>4000/μl, platelets > 100,000/μl and a hemoglobin level > 9.5 g/dl. Adequate baseline hepatic function, defined as a total bilirubin level < 2 mg/dl, SGPT and SGOT < 2.5 times the upper limits of normal. Creatinine < 1.5 mg/dl or creatinine clearance > 60 ml/min.
10. All females of childbearing potential must have a negative serum or urine pregnancy test obtained within 2 days prior to initiation of treatment and use effective contraception during the period of therapy.
11. At least one month from the last chemotherapy administration.
12. Provision of adequate paraffin-embedded tumor tissue for translational studies (optional).

Exclusion Criteria:

1. Other histological types (germ cell, granulose tumors etc)
2. History of atrial or ventricular arrhythmias and/or history of congestive heart failure, even if medically controlled. History of clinical and electrocardiographically documented myocardial infarction within the last 6 months from study entry
3. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)
4. Pre-existing motor or sensory neurotoxicity grade 2 according to the WHO criteria (intolerable paresthesia and/or marked motor loss or worse)
5. History of any treatment for CA125 relapse
6. Known, severe hypersensitivity to temsirolimus or any of the excipients of this product
7. Other coexisting malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
8. Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
9. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (eg unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
10. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2.5 times the ULRR.
11. Active infection or evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial/ receive protocol treatment
12. Concomitant use of Cyp3 A inducers (phenytoin, carbamazepine, rifampicin, barbiturates or St John's Wort) should be avoided and as should treatment with strong CyP 3A inhibitors
13. Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Clinical progression free survival. | 6-month

SECONDARY OUTCOMES:
Progression Free Survival (PFS),Survival, CA125 response rate, Safety | Duration of the study

CONTACTS AND LOCATIONS:
Locations (12):
- Greece (12):
  - "Alexandra" Hospital, Dept. of Clinical Therapeutics, Oncology, Athens
  - "Attikon" University Hospital, 2nd Dept. of Internal Medicine-Propaedeutic, Oncology Section, Athens
  - Hygeia Hospital, 1st Dept. of Medical Oncology, Athens
  - Hygeia Hospital, 2nd Dept. of Medical Oncology, Athens
  - Agii Anargiri Cancer Hospital, 3rd Dept. of Medical Oncology, Athens
  - Chania General Hospital, Oncology Dept., Chania
  - Ioannina University Hospital, Dept. of Medical Oncology, Ioannina
  - Larissa University Hospital, Oncology Dept., Larissa
  - University Hospital of Patras, Oncology Dept, Pátrai
  - Metropolitan Hospital, 1st Dept. of Medical Oncology, Pireaus
  - Metropolitan Hospital, 2nd Dept. of Medical Oncology, Pireaus
  - "Papageorgiou" General Hospital, Dept. of Medical Oncology, Thessaloniki